CLINICAL TRIAL: NCT01274806
Title: TAKE-CARE: EFFECTIVENESS OF A PHYSICAL THERAPY COMBINING CORE STABILITY EXERCISE AND MASSAGE IN CANCER RELATED SYMPTOMS
Brief Title: Take-Care Program: Effectiveness of a Physical Therapy Program on Cancer Related Symptoms
Acronym: TAKE-CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Salud Carlos III (Other Government)
Collaborators: Universidad de Granada (Other)
Responsible Party: Manuel Arroyo Morales, University of Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PI0890418; ETES0890418 (Other Grant/Funding Number: ETES0890418)
Record Dates: First submitted 2010-12-22; First posted 2011-01-12 (Estimated); Last update posted 2011-01-12 (Estimated); Status verified 2009-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; physical therapy; massage; core stability
MeSH Terms: conditions — Breast Neoplasms | interventions — Physical Therapy Modalities; Exercise; Relaxation Therapy; Post-Exercise Recovery Techniques

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual care (No Intervention)
- Physical therapy (Experimental)
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — Core Stability Exercise, Endurance training, recovery massage
  Other Names: Exercise; Relaxation techniques; Recovery techniques
  Arms: Physical therapy

SUMMARY:
Effectiveness of a physical therapy program focussed on core stability exercise and massage as a recovery method in breast cancer survivors after oncology treatment.

DETAILED DESCRIPTION:
Eligibility Criteria

1, had a diagnosis of breast cancer (stage I-IIIA); 2, between 25-65 years; 3, finished co-adjuvant treatment except hormone-therapy; 4, not having active cancer; 5, interest to improve their lifestyle increasing physical activity; and, 6, present 3 to 5 of the following physical findings, judged by the oncologist who referred the patient: neck or shoulder pain symptoms, reduced range of motion in neck- shoulder area, reduced physical capacity, any psychological problem, increased fatigue, sleep disturbances, or any problem in coping with reduced physical and psychosocial functioning.

Principal Outcomes Fatigue Score: Piper Fatigue Scale Mood State:Profile of Mood State Quality of Life: QLQ-BR23

ELIGIBILITY:
Inclusion Criteria:

* Finished oncology treatment (chemotherapy, radiation, surgery)

Exclusion Criteria:

* Other musculoskeletal conditions.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2009-01; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Fatigue Related Cancer at 6 months | Baseline, 6 months
  Piper Fatigue Scale

SECONDARY OUTCOMES:
Change from Baseline in strength at 6 months | Baseline, six months
  Leg strength, core muscles strength, arm strength
Change from Baseline in Quality of Life at 6 months | Baseline, six months
  QLQ-Br23
Change from Baseline in profile of mood state at 6 months | Baseline, six months
  Profile of Mood State

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Arroyo-Morales, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Faculty of Health Sciences, Granada, Granada, Spain